CLINICAL TRIAL: NCT07090967
Title: The Effect of the Project Planning Course on Nursing Students' Critical Thinking, Lifelong Learning, and Individual Innovativeness Skills: A Randomized Controlled Trial
Brief Title: Effect of Project Planning Course on Nursing Students' Critical Thinking, Lifelong Learning, and Innovativeness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Merve Tuncer, Assistant Professor, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2025-1
Record Dates: First submitted 2025-05-26; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Nursing Education

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Students Taking the Project Planning Course
  Interventions: Other: Project Planning Course
- Control Group (No Intervention): Students Dont Taking the Project Planning Course

INTERVENTIONS:
Other: Project Planning Course — The Project Planning Course is conducted as a two-hour theoretical class per week. This course is being introduced for the first time in the nursing faculty curriculum. The course was conducted by two faculty members, both of whom have knowledge and experience in research and project writing. Since the goal at the end of the course was for students either to carry out a research project or to apply for a patent/utility model, it was planned for 20 students to enroll; however, 19 students chose the course. The course lasted 14 weeks in total. In the first week, topics such as what a project is, its characteristics, and its components were introduced to the students. As part of the course, students were asked to brainstorm solutions for problems they encountered in clinical settings. During the first seven weeks, theoretical lectures were delivered, and during the following five weeks, students worked with their academic advisors on research projects or patent/utility model topics.
  Arms: Intervention Group

SUMMARY:
This randomized, controlled trial investigates the impact of a Project Planning Course on third-year undergraduate nursing students' critical thinking motivation, lifelong learning skills, and individual innovativeness. Participants were randomized into two groups: an intervention group receiving the Project Planning Course and a control group with no intervention. The Project Planning Course consisted of 14 weeks of theoretical and practical training, aiming to develop students' skills in research project management and patent/utility model application. Data were collected using the Critical Thinking Motivation Scale (CTMS), the Lifelong Learning Scale (LLS), and the Individual Innovativeness Scale (IIS). Statistical analysis was conducted using non-parametric tests. The study complies with ethical standards, including approval from the relevant ethics committee, and is prospectively registered at ClinicalTrials.gov.

DETAILED DESCRIPTION:
This study explores the effects of a structured Project Planning Course on the development of essential 21st-century competencies among undergraduate nursing students. Designed as a randomized controlled trial, the study involved third-year nursing students who were randomly assigned to either an intervention group, which completed a 14-week course in project planning, or a control group that received no intervention. The intervention focused on enhancing students' abilities in research planning, innovation, and intellectual property application, including patent and utility model procedures.

To assess the impact of the course, data were collected using validated instruments: the Critical Thinking Motivation Scale (CTMS), the Lifelong Learning Scale (LLS), and the Individual Innovativeness Scale (IIS). Statistical analyses were performed using non-parametric tests appropriate for the data distribution. Ethical approval was obtained from the institutional review board, and the trial was prospectively registered at ClinicalTrials.gov. This study contributes to nursing education literature by evaluating how structured project-based learning influences students' motivation, learning orientation, and innovativeness in preparation for dynamic healthcare environments.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were as follows: age ≥ 18 years, , and willing to participate in the study.

Exclusion Criteria:

* who don't want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
critical thinking | From the beginning of the term and end of the term at 14 weeks.
  Critical Thinking Motivation Scale: The CTMS is a 19-item, six-point Likert-type scale developed by Valenzuela et al. and adapted into Turkish by Dönmez and Kaya (2016). It includes five factors under two main dimensions: "expectation" and "value." Scores are calculated by averaging item responses within each subscale. The scale has a Cronbach's alpha of 0.90. Higher scores indicate greater motivation for critical thinking.
lifelong learning | From the beginning of the term and end of the term at 14 weeks.
  Lifelong Learning Scale: The LLS, developed by Wielkiewicz and Meuwissen (2014) and adapted into Turkish by Engin et al. (2017), is a 15-item, single-factor scale rated on a five-point Likert scale. Total scores range from 15 to 75, with higher scores indicating stronger lifelong learning tendencies. The scale's Cronbach's alpha is 0.86.
Individual Innovativeness | From the beginning of the term and end of the term at 14 weeks.
  Individual Innovativeness Scale:The IIS, developed by Hurt et al. (1977) and adapted into Turkish by Kılıçer and Odabaşı (2010), is a 20-item scale with four factors: Resistance to Change, Opinion Leadership, Openness to Experience, and Risk-Taking. It uses a five-point Likert scale and has a Cronbach's alpha of 0.82. Total scores classify individuals as Innovators (>80), Early Adopters (69-80), Early Majority (57-68), Late Majority (46-56), or Laggards (<46).

CONTACTS AND LOCATIONS:
Overall Officials: Merve TUNCER, Asist. Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aley M, Lee R, Wang J, Wang J, Zheng S. Project-based learning and student outcomes in health professions education: A literature review. Health Professions Education. 2023;9(3):251-266.

DOCUMENTS (1):
  • Informed Consent Form (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT07090967/ICF_000.pdf